CLINICAL TRIAL: NCT01172912
Title: Tandem High-Dose Chemotherapy (HDCT) With Peripheral-Blood Stem-Cell Rescue for Patients With Metastatic Germ-Cell Tumors Failing First-Line Treatment
Brief Title: High-Dose Chemotherapy and Stem Cell Transplant in Treating Patients With Metastatic Germ Cell Tumors That Have Not Responded to First-Line Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ITA-MIL-INT-38-10; CDR0000682204 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2010-021898-36; EU-21054
Record Dates: First submitted 2010-07-29; First posted 2010-07-30 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Brain and Central Nervous System Tumors; Extragonadal Germ Cell Tumor; Testicular Germ Cell Tumor
Keywords: recurrent extragonadal germ cell tumor; recurrent extragonadal non-seminomatous germ cell tumor; recurrent malignant testicular germ cell tumor; stage IV extragonadal non-seminomatous germ cell tumor; stage III malignant testicular germ cell tumor; recurrent extragonadal seminoma; stage IV extragonadal seminoma; testicular mature teratoma; adult central nervous system germ cell tumor; testicular immature teratoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Testicular Germ Cell Tumor; Testicular Neoplasms | interventions — Filgrastim; pegfilgrastim; Carboplatin; Cisplatin; Dexamethasone; Etoposide; Ifosfamide; Drug Therapy; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: pegfilgrastim
Drug: carboplatin
Drug: cisplatin
Drug: dexamethasone
Drug: etoposide
Drug: ifosfamide
Other: high-dose chemotherapy with autologous stem cell rescue
Other: laboratory biomarker analysis
Procedure: autologous hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. An autologous stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy.

PURPOSE: This phase II trial is studying the side effects of giving high-dose chemotherapy together with stem cell transplant and to see how well it works in treating patients with metastatic germ cell tumors that have not responded to first-line therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the efficacy of high-dose chemotherapy comprising carboplatin and etoposide (CE) in combination with autologous hematopoietic stem cell transplantation using the CE regimen as initial salvage treatment in patients with relapsed or refractory, metastatic germ cell tumors that did not respond to first-line treatment.
* To evaluate the toxicity associated with this regimen in these patients.
* To evaluate biological correlates of outcome in patients with available tissue pre- and post-treatment.

OUTLINE:

* Conventional-dose chemotherapy: Patients receive ifosfamide on days 1 and 2, followed by cisplatin and etoposide on days 3-5, and dexamethasone on days 1-5. Patients undergo leukapheresis daily for stem cell harvest. Patients also receive conventional filgrastim (G-CSF) subcutaneously (SC) once a day beginning 48 hours after completion of chemotherapy until adequate collection of stem cells are obtained. Treatment repeats every 21 days for 1 or 2 courses.
* High-dose (HD) chemotherapy: Patients receive HD carboplatin and etoposide once a day on days 1-3. Treatments repeat every 30-40 days for 2 courses.
* Autologous hematopoietic stem cell transplantation: Patients undergo reinfusion of autologous stem cells on day 6 (after HD chemotherapy on days 1-5). Patients then receive one dose of pegfilgrastim SC beginning 6 hours after completion of stem cell infusion or conventional filgrastim SC once daily beginning 4 days after completion of stem cell infusion and continuing until blood counts recover.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed germ cell tumor (GCT) based on pathologic review at INT Milan

  * Metastatic disease
  * Relapsed or refractory disease
* Prior chemotherapy treatment for GCT without a pathologic diagnosis due to unequivocal clinical evidence of GCT and an urgent need to start therapy (elevated alpha-fetoprotein [AFP] or human chorionic gonadotropin [HCG] with pattern of metastases consistent with GCT and high tumor burden) allowed
* Unequivocal progression of measurable disease, consisting of abnormalities on 2-dimensional imaging or raised tumor markers, following 1 line of cisplatin-based chemotherapy as documented by either of the following:

  * Tumor biopsy of new, growing, or unresectable lesions demonstrating viable non-teratomatous GCT (enrollment on this study for adjuvant treatment after resection of viable GCT not allowed)
  * Increasing or abnormally elevated serum tumor markers (HCG or AFP) (increasing lactate dehydrogenase [LDH] alone does not constitute progressive disease)
* Received ≥ 3 and ≤ 6, cisplatin-based chemotherapy courses as part of first-line (initial) chemotherapy and ≤ 6 cisplatin-based chemotherapy courses
* Brain metastases allowed

  * May be treated with radiotherapy and/or surgery concurrently with cisplatin, ifosfamide, and etoposide regimen

    * Radiotherapy should not be given concurrently with mobilization phase/leukapheresis and high-dose carboplatin and etoposide

PATIENT CHARACTERISTICS:

* WBC ≥ 2,000/µL
* ANC ≥ 1,500/µL
* Platelet count ≥ 100,000/µL
* Creatinine clearance ≥ 50 cc/min (unless renal dysfunction is due to tumor obstructing the ureters, in which case eligibility will be determined by the principal investigator)
* AST/ALT < 2 times upper limit of normal (ULN) (< 5 times ULN if due to hepatic metastases)
* Total bilirubin < 1.5 times ULN
* Ejection fraction ≥ 50% by echocardiogram
* Negative serology for the following infectious diseases:

  * HIV type 1 and 2
  * Hepatitis B surface antigen (active carriers)
  * Hepatitis C
  * Cytomegalovirus (serum Ag p65 ± PCR confirmation at principal investigator discretion)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior surgery
* At least 3 weeks since prior chemotherapy
* No prior high-dose chemotherapy with peripheral blood stem cell rescue
* No more than 1 prior chemotherapy regimen for metastatic disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy
Toxicity
Biological correlates of outcome

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro M. Gianni, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione Istituto Nazionale dei Tumori, Milan, Italy